CLINICAL TRIAL: NCT04425356
Title: Evaluation of the Effectiveness of a Mindfulness Coaching Program for Stress Management: A Randomized Control Trial
Brief Title: Are Mindfulness Programs in the Workplace Effective at Reducing Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American Heart Association (Other)
Collaborators: Life Cross Training (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LifeXT2019
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Mindfulness; Occupational Stress
Keywords: Resilience, Psychological; Energy Level; Empathy; Emotional Intelligence; Satisfaction with Relationships; Happiness; Sleep Quality; Physical Health; Presenteeism; Focus; Collective Efficacy; Job Satisfaction; Job Engagement
MeSH Terms: conditions — Occupational Stress; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Three experimental groups (1 from each of the 3 different implementation sites) will receive the intervention while 3 control groups will not. The control groups will be placed on a waitlist to receive the intervention once the study period is complete.
Who Masked: Investigator
Masking Description: The primary investigator and team (including those involved with the data analysis) have no knowledge of which participants were assigned to intervention or control groups. Group assignment was conducted by Life Cross Training independently of the AHA investigation team. Participants are not blinded to their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive the LifeXT program
  Interventions: Behavioral: LifeXT Program
- Control Group (No Intervention): Wait-list control group that receives the LifeXT program after the conclusion of the study

INTERVENTIONS:
Behavioral: LifeXT Program — The intervention involves participation in and completion of the 4-month LIFEXT program, including: A baseline 15-20 minute health assessment administered online, a 50 minute introductory, one-on-one telephonic coaching session, four 50 minute one-on-one telephonic coaching sessions, optional coaching session follow-up activities (such as videos, practice exercises, and reading materials), and a post-intervention 15-20 minute health assessment administered online.
  Arms: Intervention Group

SUMMARY:
The objective of this study is to determine whether a mindfulness coaching program was efficacious at reducing work stress, improving psychological and physical health outcomes, and improving work outcomes. The target population is employed adults (18 years and older) working in the industries of media, consulting, and healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Employees who are eligible to take the company's health risk assessment and/or biometric screening
* Employees who are eligible for medical health benefits

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mindfulness | Assessed at baseline
  Mindfulness is assessed using the Mindfulness Attention Awareness Scale (MAAS) consisting of 15 items. Higher scores reflect higher levels of dispositional mindfulness. The scale has been validated in college, working adult, and cancer patient populations (Brown and Ryan, 2003). The scale range was changed from 1-6 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Mindfulness | Assessed immediately post-intervention (4 moths after baseline)
  Mindfulness is assessed using the Mindfulness Attention Awareness Scale (MAAS) consisting of 15 items. Higher scores reflect higher levels of dispositional mindfulness. The scale has been validated in college, working adult, and cancer patient populations (Brown and Ryan, 2003). The scale range was changed from 1-6 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Mindfulness | Assessed at follow-up (3 months post intervention)
  Mindfulness is assessed using the Mindfulness Attention Awareness Scale (MAAS) consisting of 15 items. Higher scores reflect higher levels of dispositional mindfulness. The scale has been validated in college, working adult, and cancer patient populations (Brown and Ryan, 2003). The scale range was changed from 1-6 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Stress | Assessed at baseline
  Stress is assessed using 4 items from the 10-item Perceived Stress Scale (PSS). The PSS has demonstrated internal consistency and validity (Cohen, 1983). The PSS asks respondents to indicate how often they felt or thought a certain way during a specified time period (i.e., over the last 2 weeks). Examples of items include, "how often have you felt that you were unable to control the important things in your life," and "how often have you felt that things were going your way." The sale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment. Higher scores reflect higher levels of perceived stress.
Stress | Assessed immediately post-intervention (4 moths after baseline)
  Stress is assessed using 4 items from the 10-item Perceived Stress Scale (PSS). The PSS has demonstrated internal consistency and validity (Cohen, 1983). The PSS asks respondents to indicate how often they felt or thought a certain way during a specified time period (i.e., over the last 2 weeks). Examples of items include, "how often have you felt that you were unable to control the important things in your life," and "how often have you felt that things were going your way." The sale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment. Higher scores reflect higher levels of perceived stress.
Stress | Assessed at follow-up (3 months post intervention)
  Stress is assessed using 4 items from the 10-item Perceived Stress Scale (PSS). The PSS has demonstrated internal consistency and validity (Cohen, 1983). The PSS asks respondents to indicate how often they felt or thought a certain way during a specified time period (i.e., over the last 2 weeks). Examples of items include, "how often have you felt that you were unable to control the important things in your life," and "how often have you felt that things were going your way." The sale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment. Higher scores reflect higher levels of perceived stress.

SECONDARY OUTCOMES:
Energy | Assessed at baseline
  Energy (or vitality) is assessed using the Short-Form-36 (SP-36) which consists of 36 items to assess vitality. Higher scores reflect higher levels of vitality. The SP-36 inspired the question, "During the past month, how often did you experience the following?" in the LIFE XT assessment. The questionnaire asks this question about four items: felt full of pep, felt tired, had a lot energy and felt worn out. Each of these questions is on a scale from 1-7, for a total of 28 points and a higher score reflecting higher energy levels.
Energy | Assessed immediately post-intervention (4 months after baseline)
  Energy (or vitality) is assessed using the Short-Form-36 (SP-36) which consists of 36 items to assess vitality. Higher scores reflect higher levels of vitality. The SP-36 inspired the question, "During the past month, how often did you experience the following?" in the LIFE XT assessment. The questionnaire asks this question about four items: felt full of pep, felt tired, had a lot energy and felt worn out. Each of these questions is on a scale from 1-7, for a total of 28 points and a higher score reflecting higher energy levels.
Energy | Assessed at follow-up (3 months post intervention)
  Energy (or vitality) is assessed using the Short-Form-36 (SP-36) which consists of 36 items to assess vitality. Higher scores reflect higher levels of vitality. The SP-36 inspired the question, "During the past month, how often did you experience the following?" in the LIFE XT assessment. The questionnaire asks this question about four items: felt full of pep, felt tired, had a lot energy and felt worn out. Each of these questions is on a scale from 1-7, for a total of 28 points and a higher score reflecting higher energy levels.
Empathy | Assessed at baseline
  Empathy is assessed using the Empathic Concern subscale of the Interpersonal Reactivity Index developed by Davis (1980). The subscale includes 4 items. Examples of items include, "I often have tender, concerned feelings for people less fortunate than I am" and "Other people's misfortunes do not usually disturb me a great deal." The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Empathy | Assessed immediately post-intervention (4 months after baseline)
  Empathy is assessed using the Empathic Concern subscale of the Interpersonal Reactivity Index developed by Davis (1980). The subscale includes 4 items. Examples of items include, "I often have tender, concerned feelings for people less fortunate than I am" and "Other people's misfortunes do not usually disturb me a great deal." The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Empathy | Assessed at follow-up (3 months post intervention)
  Empathy is assessed using the Empathic Concern subscale of the Interpersonal Reactivity Index developed by Davis (1980). The subscale includes 4 items. Examples of items include, "I often have tender, concerned feelings for people less fortunate than I am" and "Other people's misfortunes do not usually disturb me a great deal." The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Emotional Health | Assessed at baseline
  Emotional health is assessed using 1 question, "How would you rate your emotional health overall during the past month?" The question was developed by the LIFE XT personal health assessment author.
Emotional Health | Assessed immediately post-intervention (4 months after baseline)
  Emotional health is assessed using 1 question, "How would you rate your emotional health overall during the past month?" The question was developed by the LIFE XT personal health assessment author.
Emotional Health | Assessed at follow-up (3 months post intervention)
  Emotional health is assessed using 1 question, "How would you rate your emotional health overall during the past month?" The question was developed by the LIFE XT personal health assessment author.
Relationships (Satisfaction with): questionnaire | Assessed at baseline
  Satisfaction in relationships with children, parents, friends, and relatives is assessed with 4 items, one for each relationship domain. For each of the four relationship domains, the question asks, "On average, how satisfied are you in your relationship with your [parents/friends/relatives]". The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Relationships (Satisfaction with): questionnaire | Assessed immediately post-intervention (4 months after baseline)
  Satisfaction in relationships with children, parents, friends, and relatives is assessed with 4 items, one for each relationship domain. For each of the four relationship domains, the question asks, "On average, how satisfied are you in your relationship with your [parents/friends/relatives]". The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Relationships (Satisfaction with): questionnaire | Assessed at follow-up (3 months post intervention)
  Satisfaction in relationships with children, parents, friends, and relatives is assessed with 4 items, one for each relationship domain. For each of the four relationship domains, the question asks, "On average, how satisfied are you in your relationship with your [parents/friends/relatives]". The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Happiness (Life Satisfaction): questionnaire | Assessed at baseline
  Happiness is assessed using 5 items from the Satisfaction with Life Scale (SWLS) developed by Diener et al. The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Happiness (Life Satisfaction): questionnaire | Assessed immediately post-intervention (4 months after baseline)
  Happiness is assessed using 5 items from the Satisfaction with Life Scale (SWLS) developed by Diener et al. The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Happiness (Life Satisfaction): questionnaire | Assessed at follow-up (3 months post intervention)
  Happiness is assessed using 5 items from the Satisfaction with Life Scale (SWLS) developed by Diener et al. The scale range was changed from 1-5 to 1-7 when adapted and added into the LIFE XT personal health assessment.
Physical Health | Assessed at baseline
  Physical Health is assessed using 2 questions. The first item is based on a question developed by researchers Lorig et al., "In general, would you say your health is:… (Circle one) (Excellent = 1, Very Good = 2, Good = 3, Fair = 4, Poor = 5.)" The second question, "How would you rate your physical health overall during the past month?" was developed by the LIFE XT personal health assessment author.
Physical Health | Assessed immediately post-intervention (4 months after baseline)
  Physical Health is assessed using 2 questions. The first item is based on a question developed by researchers Lorig et al., "In general, would you say your health is:… (Circle one) (Excellent = 1, Very Good = 2, Good = 3, Fair = 4, Poor = 5.)" The second question, "How would you rate your physical health overall during the past month?" was developed by the LIFE XT personal health assessment author.
Physical Health | Assessed at follow-up (3 months post intervention)
  Physical Health is assessed using 2 questions. The first item is based on a question developed by researchers Lorig et al., "In general, would you say your health is:… (Circle one) (Excellent = 1, Very Good = 2, Good = 3, Fair = 4, Poor = 5.)" The second question, "How would you rate your physical health overall during the past month?" was developed by the LIFE XT personal health assessment author.
Sleep Quality: PSQI | Assessed at baseline
  Sleep is assessed using 1 item from the Pittsburgh Sleep Quality Index (PSQI). The item, "During the past work week, how would you rate your sleep quality overall?" assesses sleep quality. The scale range was change from very good, fairly good, fairly bad, and very bad to 1-7, where 1 is labeled poor, and 7 is labeled excellent.
Sleep Quality: PSQI | Assessed immediately post-intervention (4 months after baseline)
  Sleep is assessed using 1 item from the Pittsburgh Sleep Quality Index (PSQI). The item, "During the past work week, how would you rate your sleep quality overall?" assesses sleep quality. The scale range was change from very good, fairly good, fairly bad, and very bad to 1-7, where 1 is labeled poor, and 7 is labeled excellent.
Sleep Quality: PSQI | Assessed at follow-up (3 months post intervention)
  Sleep is assessed using 1 item from the Pittsburgh Sleep Quality Index (PSQI). The item, "During the past work week, how would you rate your sleep quality overall?" assesses sleep quality. The scale range was change from very good, fairly good, fairly bad, and very bad to 1-7, where 1 is labeled poor, and 7 is labeled excellent.
Productivity (or work impairment) | Assessed at baseline
  Work impairment is assessed using the Lam Employment Absence and Productivity Scale (LEAPS) which consists of 7 items that describe how patients are functioning at work. Higher scores indicate higher levels of work impairment. A low score reflects minimal to no work impairment. This tool has been used to help physicians make management decisions such as whether or not a patient should stay at work, whether work functioning improves along with symptoms, and whether changes in treatment are needed to optimize work functioning. It has been validated in patients with major depressive disorder (Lam et al.). The scale range was changed from 0-4
Productivity (or work impairment) | Assessed immediately post-intervention (4 months after baseline)
  Work impairment is assessed using the Lam Employment Absence and Productivity Scale (LEAPS) which consists of 7 items that describe how patients are functioning at work. Higher scores indicate higher levels of work impairment. A low score reflects minimal to no work impairment. This tool has been used to help physicians make management decisions such as whether or not a patient should stay at work, whether work functioning improves along with symptoms, and whether changes in treatment are needed to optimize work functioning. It has been validated in patients with major depressive disorder (Lam et al.). The scale range was changed from 0-4
Productivity (or work impairment) | Assessed at follow-up (3 months post intervention)
  Work impairment is assessed using the Lam Employment Absence and Productivity Scale (LEAPS) which consists of 7 items that describe how patients are functioning at work. Higher scores indicate higher levels of work impairment. A low score reflects minimal to no work impairment. This tool has been used to help physicians make management decisions such as whether or not a patient should stay at work, whether work functioning improves along with symptoms, and whether changes in treatment are needed to optimize work functioning. It has been validated in patients with major depressive disorder (Lam et al.). The scale range was changed from 0-4
Presenteeism | Assessed at baseline
  Presenteeism is measured using 5 items from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The items reflect what an employee may do or feel at work.
Presenteeism | Assessed immediately post-intervention (4 months after baseline)
  Presenteeism is measured using 5 items from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The items reflect what an employee may do or feel at work.
Presenteeism | Assessed at follow-up (3 months post intervention)
  Presenteeism is measured using 5 items from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The items reflect what an employee may do or feel at work.
Employee Retention | Assessed at baseline
  Employee Retention is measured using 1 item from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The question is, "How likely are you, currently, to consider leaving your job due to work related stress?"
Employee Retention | Assessed immediately post-intervention (4 months after baseline)
  Employee Retention is measured using 1 item from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The question is, "How likely are you, currently, to consider leaving your job due to work related stress?"
Employee Retention | Assessed at follow-up (3 months post intervention)
  Employee Retention is measured using 1 item from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The question is, "How likely are you, currently, to consider leaving your job due to work related stress?"
Teamwork (collective efficacy) | Assessed at baseline
  Collective efficacy, or people's shared beliefs in their collective capacity to achieve desired outcomes, is assessed using 5 items adapted from the family efficacy scale for soldiers (Bandura, 2006). These items were adapted in the LIFE XT personal health assessment for employees to reflect their confidence in their work teams.
Teamwork (collective efficacy) | Assessed immediately post-intervention (4 months after baseline)
  Collective efficacy, or people's shared beliefs in their collective capacity to achieve desired outcomes, is assessed using 5 items adapted from the family efficacy scale for soldiers (Bandura, 2006). These items were adapted in the LIFE XT personal health assessment for employees to reflect their confidence in their work teams.
Teamwork (collective efficacy) | Assessed at follow-up (3 months post intervention)
  Collective efficacy, or people's shared beliefs in their collective capacity to achieve desired outcomes, is assessed using 5 items adapted from the family efficacy scale for soldiers (Bandura, 2006). These items were adapted in the LIFE XT personal health assessment for employees to reflect their confidence in their work teams.
Job Satisfaction: WOS | Assessed at baseline
  Job satisfaction is measured using 5 items from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The items describe how an individual feels about their work. The items use a scale from strongly disagree to strongly agree.
Job Satisfaction: WOS | Assessed immediately post-intervention (4 months after baseline)
  Job satisfaction is measured using 5 items from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The items describe how an individual feels about their work. The items use a scale from strongly disagree to strongly agree.
Job Satisfaction: WOS | Assessed at follow-up (3 months post intervention)
  Job satisfaction is measured using 5 items from the Workplace Outcome Suite (WOS) instrument developed by Chestnut Global Partners, a provider of employee assistance programs. The items describe how an individual feels about their work. The items use a scale from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Calitz, MPP, Principal Investigator — American Heart Association
Locations (3):
- United States (3):
  - Navicent Health, Macon, Georgia
  - Spark Foundry, Chicago, Illinois
  - The Leo Burnett Media Agency, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No